CLINICAL TRIAL: NCT03476915
Title: Incidence of Developmental Hip Dysplasia by Ultrasonographic Screening of Asymptomatic Infants Less Than 6 Months Old at Assiut University Hospital Outpatient Clinics
Brief Title: Developmental Hip Dysplasia by Ultrasonographic Screening of Asymptomatic Infants at Assiut University Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sondos Hassan, principal investigator, Assiut University
Other Study IDs: DHD2017
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- screened infants: Asymptomatic infants under age of 6 months, presenting to the pediatric orthopaedic outpatient clinic at Assiut university hospital for other problems will be subjected to ultrasound examination of the hip joint.
  Interventions: Other: ultrasound examination of the hip joint

INTERVENTIONS:
Other: ultrasound examination of the hip joint — US examination by US machine , Midray model DP-2200 made in China , with a high frequency (5-10 MHZ) linear transducer using the previously described Graf method for assessment of both hip joints.

SUMMARY:
Developmental dysplasia of the hip (DDH), formerly known as congenital dislocation of the hip, comprises a spectrum of abnormalities that include abnormal acetabular shape (dysplasia) and malposition of the femoral head.

DETAILED DESCRIPTION:
The origin and pathogenesis of DDH are multifactorial. Abnormal laxity of the ligaments and hip capsule is seen in patients with DDH. The maternal hormone relaxin may also be a factor. Extreme hip flexion with knee extension, as in the breech position, tends to promote femoral head dislocation and leads to the shortening and contracture of the iliopsoas muscle.

It was previously reported that DDH was the underlying aetiology in about 25 % of the performed hip replacements under the age of 40 years and the initial diagnosis age ranged from 0 to 39 years, with a mean of 8 years in these patients.

The main purpose of a newborn hip screening program is to detect DDH as early as possible, so that early treatment can be given and the need for surgical treatment as well as the development of residual hip dysplasia can be avoided.

Ultrasonography offers distinct advantages compared with other imaging techniques: unlike plain radiography, it can distinguish the cartilaginous components of the acetabulum and the femoral head from other soft tissue structures, real-time US permits multiplanar examinations that can early determine the position of the femoral head in respect to the acetabulum; thus it provides the same type of information that can be obtained with arthrography, computerized tomography, or magnetic resonance imaging, but at lower cost, although ultrasonography is more expensive than plain radiography, it doesn't require sedation and doesn't involve ionizing radiation, unlike other techniques and it allows observation of changes in hip position with movement.

ELIGIBILITY:
Inclusion Criteria:

* All infants under the age of 6 months attending Pediatric Orthopedic outpatient clinics at Assiut university hospital in the period between 1st of January 2017 to 30th of December 2017.

Exclusion Criteria:

* Age older than 6 months
* Having any hip joint complaints

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants under the age of 6 months attending Pediatric Orthopedic outpatient clinics at Assiut university hospital in the period between 1st of January 2017 to 30th of December 2017.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
The alpha and the beta angels of the hip by ultrasound | baseline
  The α-angle is a measure of acetabular depth and is the angle formed between the acetabular roof and vertical cortex of the ilium. The beta angle is the angle formed between the vertical cortex of the ilium and triangular labral fibrocartilage, It represents the acetabular cartilaginous roof modeling

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dezateux C, Rosendahl K. Developmental dysplasia of the hip. Lancet. 2007 May 5;369(9572):1541-1552. doi: 10.1016/S0140-6736(07)60710-7. PMID 17482986
- [Background] Engesaeter IO, Lehmann T, Laborie LB, Lie SA, Rosendahl K, Engesaeter LB. Total hip replacement in young adults with hip dysplasia: age at diagnosis, previous treatment, quality of life, and validation of diagnoses reported to the Norwegian Arthroplasty Register between 1987 and 2007. Acta Orthop. 2011 Apr;82(2):149-54. doi: 10.3109/17453674.2011.566146. Epub 2011 Mar 24. PMID 21434808
- [Background] Sewell MD, Rosendahl K, Eastwood DM. Developmental dysplasia of the hip. BMJ. 2009 Nov 24;339:b4454. doi: 10.1136/bmj.b4454. No abstract available. PMID 19934187
- [Background] Wientroub S, Grill F. Ultrasonography in developmental dysplasia of the hip. J Bone Joint Surg Am. 2000 Jul;82-A(7):1004-18. doi: 10.2106/00004623-200007000-00012. No abstract available. PMID 10901315